CLINICAL TRIAL: NCT03151655
Title: Changing Opioid Users' Negative Attitudes Toward Medication Assisted Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not secured for the project as expected, so we were unable to proceed with the project.
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Brandon Gaudiano, Multiple Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1610-001
Record Dates: First submitted 2016-10-14; First posted 2017-05-12 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MATTeRS Video (Experimental)
  Interventions: Behavioral: MATTeRS Video
- Didactic Video (Active Comparator)
  Interventions: Behavioral: Didactic Video

INTERVENTIONS:
Behavioral: MATTeRS Video — Narrative-based video intervention and accompanying workbook
  Arms: MATTeRS Video
Behavioral: Didactic Video — Education only video
  Arms: Didactic Video

SUMMARY:
In this treatment development project, the investigators propose to develop and assess the feasibility and acceptability of a narrative-based video intervention and accompanying workbook (entitled MATTeRS: Medication Assisted Treatments: Telling Real Stories) designed to be used by people in inpatient opioid detoxification. Using the Health Belief Model as a framework, videos will provide information about the uses and outcomes of Medication Assisted Treatments (MATs) compared to other or no post-detoxification treatment through the use of narratives from real people's lives.

ELIGIBILITY:
Inclusion Criteria:

1. Currently undergoing inpatient opioid detoxification;
2. Qualify for use of one or more MATs;
3. Have health insurance;
4. Able to read and speak English;
5. Aged 18 or older;
6. No suicide ideation or behavior requiring immediate attention;
7. Live in the Rhode Island or Massachusetts area and have a working telephone;
8. Able to provide two contact persons to verify location and in case we are unable to reach the participant during the study;
9. Do not have probation/parole requirements that might interfere with protocol participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Initiation of Medication Assisted Treatment | 1 Month Post-Discharge
  Whether or not patients started medication-assisted treatment during the assessment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No